CLINICAL TRIAL: NCT01279798
Title: Expanded Access Multicenter Study of Lucanix® (Belagenpumatucel-L) in Advanced Non-small Cell Lung Cancer.
Brief Title: Expanded Access Multicenter Study of Lucanix® (Belagenpumatucel-L)
Status: No longer available | Type: Expanded Access
Sponsor: NovaRx Corporation (Industry)
Responsible Party: Habib Fakhrai, PhD, Chief Scientific Officer and Executive Vice Chairman of the Board, NovaRx Corporation
Other Study IDs: NR001-04
Record Dates: First submitted 2010-10-29; First posted 2011-01-19 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Cancer; NSCLC; stage III or IV NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — belagenpumatucel L

INTERVENTIONS:
Biological: Lucanix® (belagenpumatucel-L) — Subjects will receive up to 12 monthly (28-35 day interval) Lucanix injections at a dose of 2.5 × 10e7 cells per injection.
  Other Names: Lucanix

SUMMARY:
This is an expanded access protocol designed to make Lucanix® available to subjects with advanced non-small cell lung cancer (NSCLC) who are not eligible for the Phase III Protocol, NR001-03. A total of 45 patients will be enrolled into the study.

DETAILED DESCRIPTION:
The primary objective of this study is to increase the overall survival of the study subjects by providing expanded access to Lucanix. Overall survival and progression-free survivals will be compared with historical controls.

The secondary objectives of this study are:

* Evaluate the best overall tumor response.
* Evaluate progression-free survival (PFS).
* Evaluate treatment toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* ≥ 18 years
* Histological confirmed non-curable stage III or IV NSCLC.
* Must have completed at least one (1) regimen of anti-cancer therapy.
* Following frontline therapy, subjects must observe the following wash- out periods:

  * Subjects with stable disease or better must have received the last anti-cancer therapy not less than five months prior to enrollment.
  * Subjects with progressive disease must have received the last anti-cancer therapy at least one (1) month prior to enrollment.
* All subjects who have received two (2) or more regimens of therapy must have received the last anti-cancer therapy at least one (1) month prior to enrollment.
* Performance status (ECOG) ≤ 2
* Absolute granulocyte count ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Total Bilirubin ≤ 2× Upper Limit of Normal
* AST and ALT ≤ 2× Upper Limit of Normal
* Creatinine ≤ 2× Upper Limit of Normal
* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Concurrent systemic steroids > 2 mg prednisone/day
* Prior splenectomy
* Any chemotherapy, steroid therapy, or investigational anti-cancer agent within 4 weeks of study entry.
* Subjects who received prior monotherapy with Lucanix.
* Symptomatic brain metastases unless treated and stable for ≥ 2 months
* Known HIV positivity
* Serious non-malignant disease (e.g., congestive heart failure, or active uncontrolled bacterial, viral, or fungal infections), or other conditions which, in the opinion of the investigator would compromise protocol objectives.
* Prior malignancy (excluding non-melanoma carcinomas of the skin) unless in remission for ≥ 2 years
* History of psychiatric disorder that would impede adherence to protocol
* Pregnant or nursing women or refusal to practice contraception if of reproductive potential

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Innovative Research Center of California, San Diego, California, United States

REFERENCES:
- [Result] Nemunaitis J, Dillman RO, Schwarzenberger PO, Senzer N, Cunningham C, Cutler J, Tong A, Kumar P, Pappen B, Hamilton C, DeVol E, Maples PB, Liu L, Chamberlin T, Shawler DL, Fakhrai H. Phase II study of belagenpumatucel-L, a transforming growth factor beta-2 antisense gene-modified allogeneic tumor cell vaccine in non-small-cell lung cancer. J Clin Oncol. 2006 Oct 10;24(29):4721-30. doi: 10.1200/JCO.2005.05.5335. Epub 2006 Sep 11. PMID 16966690
- See also: NovaRx Website — http://www.novarx.com/